CLINICAL TRIAL: NCT06651645
Title: Pre- vs Post-COVID-19 Pandemic Risk-adjusted Survival Rates in the US Hospitals: Retrospective Cohort Study of Hospital Performance
Brief Title: Pre- vs Post-Pandemic Risk-adjusted Survival Rates in the US Hospitals
Status: Active, not recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Sameer Kadri, M.D., Tenure Track Investigator, National Institutes of Health Clinical Center (CC)
Other Study IDs: BD022390
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-10

CONDITIONS: In-hospital Mortality; Non-COVID Deaths; Surge
Keywords: In-hospital mortality; Post pandemic hospital performance; Surge; Hospital recovery; Hospital performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Pre-pandemic admissions: Patients admitted between January 1, 2018 - February 29, 2020 with one of the following five primary diagnoses of acute myocardial infarction, stroke, heart failure, pneumonia, and chronic obstructive pulmonary disease in alignment with the Centers for Medicare and Medicaid Service's (CMS's) condition-specific mortality measures reporting
- Post-pandemic admissions: Patients admitted between May 1, 2022 and May 31, 2023 without a diagnosis for COVID-19 and with one of the following five primary diagnoses of acute myocardial infarction, stroke, heart failure, pneumonia, and chronic obstructive pulmonary disease in alignment with the Centers for Medicare and Medicaid Service's (CMS's) condition-specific mortality measures reporting.
  Interventions: Other: COVID-19 Surge
- Pandemic admissions: Patients admitted between March 1, 2020 and April 30, 2022 without a diagnosis for COVID-19 and with one of the following five primary diagnoses of acute myocardial infarction, stroke, heart failure, pneumonia, and chronic obstructive pulmonary disease in alignment with the Centers for Medicare and Medicaid Service's (CMS's) condition-specific mortality measures reporting
  Interventions: Other: COVID-19 Surge

INTERVENTIONS:
Other: COVID-19 Surge — Impact of COVID-19 pandemic on hospital care delivery
  Groups: Pandemic admissions; Post-pandemic admissions

SUMMARY:
This study aims to perform a retrospective cohort study of administrative health data to understand how care delivery performance varies across US hospitals post-COVID-19 pandemic compared to the pre-pandemic performance. We also hope to identify which factors contribute to performance changes.

ELIGIBILITY:
The study cohort will include one random encounter per patient for all adult (age ≥18years) encounters. All inpatients with the Premier healthcare database (PINC-AI) and those patients who were admitted under observation status and expired in the hospital or those who presented acutely to the emergency department and died in the emergency department will be considered as inpatients for the purpose of this study as per prior precedence in including such patients.

All pediatric inpatients, skilled nursing facilities inpatients, long term acute care inpatients, rehabilitation facility inpatients, psychiatric inpatients, hospice inpatients, chemical dependency unit inpatients and deceased organ donor inpatients are excluded after applying encounter level exclusion criteria from this inpatient cohort. Application of this encounter level exclusion will also preferentially exclude any children hospitals, skilled nursing facilities, acute long term care facilities, psychiatry hospitals, inpatient hospices and chemical dependency units.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients admitted to a hospital represented with the PINC-AI hospital database.
Sampling Method: Non-Probability Sample
Enrollment: 30000000 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Adjusted in-hospital mortality | During hospital admission
  Our primary outcome will be based on a composite measure of in-hospital mortality or discharge to hospice as determined by discharge status code. The primary outcome will itself be expressed as a modified standardized mortality ration (mSMR) calculated as mean-shrunken number of observed deaths or discharge to hospice divided by the expected number of deaths or discharge to hospice for a center in that post-pandemic month assuming the effects of a typical center in the pre-pandemic era.

SECONDARY OUTCOMES:
Rates of potential inpatient complications (PICs) | During hospital admission
  PICs are complications developed during the hospital stay which may reflect the performance changes post pandemic due to circumstances observed during the pandemic. List of PICs will be curated as has been done previously using Premier Healthcare Database as reported in Korvink et al. Med Care, 2023. For each of the patient, we will calculate the cumulative number of PICs developed during their inpatient stay, which would be a sum of individual counts of PICs out of the list of 74 total possible PICs. Eventually, observed and expected rate of PICs normalized to the length of stay will be calculated with analysis restricted to within hospitals after adjusting for patient level covariates. Subsequently, risk factor model will include hospital level factors to assess association of these factors to aggregate rates of PICs in the cohort to identify factors associated with better or poor performance post pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Maniraj Neupane, MD, Ph.D., Principal Investigator — Grand Island Regional Medical Center
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No